CLINICAL TRIAL: NCT07149805
Title: Surgery Improves Survival Rate in Patients With Takayasu Arteritis: a Retrospective Observational Study
Brief Title: Surgery Benefits Takayasu Arteritis With Stenosis in the Descending Aorta
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Yuexin Chen, professor, Peking Union Medical College Hospital
Other Study IDs: 2022-PUMCH-A-191; BJZQ2024001 (Other Grant/Funding Number: The Education Committee of Beijing); UBJ06532 (Other Grant/Funding Number: National Health Commission of the People's Republic of China)
Record Dates: First submitted 2025-07-18; First posted 2025-09-02 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-07

CONDITIONS: Takayasu Arteritis
MeSH Terms: conditions — Takayasu Arteritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- surgerical group: Patients who underwent surgical treatment
  Interventions: Procedure: open surgery or interventional treatment
- conservative group: Patients who underwent conservative treatment

INTERVENTIONS:
Procedure: open surgery or interventional treatment — open surgery or interventional treatment
  Groups: surgerical group

SUMMARY:
The long-term prognosis and optimal management for Takayasu arteritis(TA) patients with severe stenosis of the descending thoracic and abdominal aorta remain undefined. We want to compare the clinical outcomes of surgical intervention and medical management.

ELIGIBILITY:
Inclusion Criteria:

1. fulfilling the 1990 American College of Rheumatology criteria for the diagnosis of TA;
2. having at least one site with severe narrowing in the descending thoracic and abdominal aorta;
3. having symptoms caused by TA-related stenosis, such as uncontrolled hypertension, heart failure, renal ischemia, dizziness, visual disturbances, and claudication

Exclusion Criteria:

Patients with arterial stenosis due to other reasons (such as typical atherosclerosis, congenital coarctation of the aorta, and anatomical abnormality) were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: inpatients at Peking Union Medical College Hospital
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
all-cause mortality rate | Patients underwent follow-up from discharge until study termination (3 years to 11 years) or death, whichever came first
all-cause mortality rate | Patients underwent follow-up from discharge (3 years to 11 years) until study termination or death, whichever came first

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD